CLINICAL TRIAL: NCT00391911
Title: A Randomized Factorial Trial of N-Acetylcysteine and Continuous Veno-Venous Hemo(Dia)Filtration for Rhabdomyolysis
Brief Title: Study of N-Acetylcysteine (NAC) and Continuous Renal Replacement Therapy (CRRT) for the Treatment of Rhabdomyolysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Alexandra Hospital (Other)
Collaborators: University of Alberta (Other); Gambro Renal Products, Inc. (Industry)
Responsible Party: Principal Investigator, Demetrios J. Kutsogiannis, MD MHS FRCPC, Royal Alexandra Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RHABDO 2006; Health Canada Control # 108739 (Other: Health Canada)
Record Dates: First submitted 2006-10-24; First posted 2006-10-25 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Rhabdomyolysis
Keywords: Rhabdomyolysis; CRRT; N-Acetylcysteine
MeSH Terms: conditions — Rhabdomyolysis | interventions — Acetylcysteine; N-monoacetylcystine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- NAC and CRRT (Active Comparator): N-Acetylcysteine and CRRT Patients are assigned to N-Acetylcysteine and CRRT. The N-Acetylcysteine is blinded to everyone except pharmacy. The CRRT is open label,
  Interventions: Drug: N-Acetylcysteine
- NAC and non CRRT (Other): Patients are assigned to N-Acetylcysteine and CRRT. The N-Acetylcysteine is blinded to everyone except pharmacy. The CRRT is open label as would be impossible to blind
  Interventions: Other: N-Acetylcystine and Non CRRT
- Placebo and CRRT (Other): Patients are assigned to placebo treatment and CRRT. The N-Acetylcysteine/placebo is blinded to everyone except pharmacy. The CRRT is open label.
  Interventions: Other: Placebo and CRRT
- Placebo and Non CRRT (Other): Patients are assigned to Placebo and non-CRRT. This is the standard of care arm. The N-Acetylcysteine/placebo is blinded to everyone except pharmacy. The CRRT/non CRRT is open label as would be impossible to blind
  Interventions: Other: Placebo and Non CRRT

INTERVENTIONS:
Drug: N-Acetylcysteine — Patients are assigned to either N-Acetylcysteine or placebo. Dose is weight based Placebo is normal saline or D5W
  Other Names: NAC
  Arms: NAC and CRRT
Other: N-Acetylcystine and Non CRRT — Patients are assigned to N-Acetylcysteine and CRRT. The N-Acetylcysteine is blinded to everyone except pharmacy. The CRRT is open label as would be impossible to blind
  Other Names: NAC only
  Arms: NAC and non CRRT
Other: Placebo and CRRT — Patients are assigned to Placebo and CRRT. The N-Acetylcysteine/Placebo is blinded to everyone except pharmacy. The CRRT is open label
  Other Names: Placebo
  Arms: Placebo and CRRT
Other: Placebo and Non CRRT — Patients are assigned to Placebo and non-CRRT. The N-Acetylcysteine/placebo is blinded to everyone except pharmacy. The CRRT/non CRRT is open label as would be impossible to blind
  Other Names: Placebo - no CRRT
  Arms: Placebo and Non CRRT

SUMMARY:
Rhabdomyolysis has many causes including trauma, muscle crush injuries, lack of blood supply to an arm or leg, burns, seizures, drugs and hereditary disorders. Rhabdomyolysis causes the breakdown of muscle cells and the release of a molecule called myoglobin. Myoglobin is very harmful to the kidneys and can lead to kidney failure.

Continuous dialysis has been shown to remove the myoglobin molecule from the blood in patients with rhabdomyolysis. N-Acetylcysteine (NAC) has been used in patients receiving contrast dye for x-rays and has shown less worsening of kidney function compared to patients not receiving NAC.

Early and aggressive treatment of patients with rhabdomyolysis with standard therapy, continuous dialysis and a drug called N-acetylcysteine (NAC) may prevent the development of acute kidney failure. Patients who develop kidney failure from this disorder are often critically ill and have a much higher chance of not surviving than those who do not develop kidney failure.

The purpose of this study is to determine if the use of NAC and Continuous Veno-Venous hemo(dia)filtration (CRRT)early in the course of rhabdomyolysis (in addition to standard therapy)decreases the chance of developing acute renal failure

DETAILED DESCRIPTION:
Rhabdomyolysis may be defined as a clinical or biochemical syndrome which may result from a large variety of diseases, trauma, or toxic insults to skeletal muscle. The damage to the integrity of the sarcolemma of skeletal muscle leads to the release of potentially toxic muscle cell components into the circulation, specifically myoglobin into the plasma.

The three main principals of therapy for myoglobinuric renal failure include 1) correction of hypovolemia/ renal ischemia, 2) increase the clearance of heme proteins from both the circulation and the kidneys, 3) attenuate the adverse effects of heme proteins on the proximal tubule epithelium. Consequently, therapy for rhabdomyolysis is limited to aggressive rehydration with Ringer's lactate or normal saline, forced diuresis with mannitol, and urinary alkalinization with intravenous bicarbonate.

Hypothesis

1. The use of N-acetylcysteine (NAC) and continuous veno-venous hemo(dia)filtration (CRRT) early in the course of rhabdomyolysis as an adjunct to 'standard therapy' (rehydration, mannitol diuresis, systemic alkalinization) respectively decreases the nephrotoxicity and improves elimination of systemic myoglobin. Consequently both therapies independently prevent the deterioration of renal glomerular and tubular function and establishment of acute renal failure.
2. There exists a positive interaction between the use of N-acetylcysteine and CRRT in the prevention of acute renal failure secondary to rhabdomyolysis.

Objectives Primary objective is to compare creatinine and myoglobin clearance as well as the glomerular filtration rate over the course of 192 hours in patients with rhabdomyolysis treated with NAC, early CRRT, both CRRT and NAC or neither of the two therapies. Secondary objectives are to : 1) Compare excretion of urine B-NAG, B1-macroglobulin, and microalbumin, as indicators of renal tubular and glomerular damage over the course of 192 hours in subjects with rhabdomyolysis treated with NAC, early CRRT, both therapies, or neither therapies 2) To compare ICU and hospital mortality and length of stay as well as the proportion of subjects with recovery of renal function at 14 and 28 days following randomization in patients with rhabdomyolysis treated with NAC, early CRRT, both therapies, or neither therapies 3) To determine clinical and biochemical risk factors for renal failure development in subjects with rhabdomyolysis.

ELIGIBILITY:
Inclusion Criteria:

1. Randomization within 96 hours of medical or surgical diagnosis consistent with rhabdomyolysis
2. >18 yrs old
3. Meeting any one of the following (estimated ARF risk >20% )

   * CK >25,000 IU/L
   * Injury Severity Score >16 and CK >5000 IU/L
   * Age >55 and CK >5000 IU/L
4. Clinical suspicion of high probability of developing acute renal failure
5. Informed consent

Exclusion Criteria:

1. Allergic reaction to N-acetylcysteine.
2. Previous wish not to include dialysis as part of medical therapy.
3. Clinical and biochemical indications for dialysis or ultrafiltration at the time of screening:

   * Massive fluid overload unresponsive to diuretics and requiring ultrafiltration.
   * Refractory acidosis with a persistent serum pH < 7.20 despite HCO3 therapy.
   * Hyperkalemia with EKG changes necessitating dialysis for the removal of potassium.
   * Pericardial friction rub from uremic pericarditis.
4. RIFLE category Failure defined by one of:

   * Increase serum creatinine x 3, GFR decrease 75% OR
   * SCreat ≥ 4mg/dl (354 umol/L) (acute rise ≥ 0.5mg/dl [44 umol/L])
   * UO < 0.3ml/kg/h x 24h or anuria x 12 hours
5. RIFLE category Loss - persistent ARF =complete loss of kidney function > 4 weeks
6. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures include serial measurements of markers of renal glomerular function and damage and markers of renal tubular function and damage | day 1-28

SECONDARY OUTCOMES:
Secondary outcome measures include all-cause ICU mortality and hospital mortality, ICU and hospital length of stay. | ICU admission until hospital discharge
Renal specific outcomes will include the development of Renal Failure, Loss or End Stage Kidney Disease based on the RIFLE classification system. | at day 28

CONTACTS AND LOCATIONS:
Overall Officials: Demetrios J. Kutsogiannis, M.D., Principal Investigator — University of Alberta
Locations (2):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada
- King Fahad National Guard Hospital, Riyadh, Saudi Arabia

REFERENCES:
- [Background] Abul-Ezz SR, Walker PD, Shah SV. Role of glutathione in an animal model of myoglobinuric acute renal failure. Proc Natl Acad Sci U S A. 1991 Nov 1;88(21):9833-7. doi: 10.1073/pnas.88.21.9833. PMID 1946409
- [Background] Tepel M, van der Giet M, Schwarzfeld C, Laufer U, Liermann D, Zidek W. Prevention of radiographic-contrast-agent-induced reductions in renal function by acetylcysteine. N Engl J Med. 2000 Jul 20;343(3):180-4. doi: 10.1056/NEJM200007203430304. PMID 10900277
- [Background] Briguori C, Manganelli F, Scarpato P, Elia PP, Golia B, Riviezzo G, Lepore S, Librera M, Villari B, Colombo A, Ricciardelli B. Acetylcysteine and contrast agent-associated nephrotoxicity. J Am Coll Cardiol. 2002 Jul 17;40(2):298-303. doi: 10.1016/s0735-1097(02)01958-7. PMID 12106935
- [Background] Sochman J. N-acetylcysteine in acute cardiology: 10 years later: what do we know and what would we like to know?! J Am Coll Cardiol. 2002 May 1;39(9):1422-8. doi: 10.1016/s0735-1097(02)01797-7. PMID 11985902
- [Background] Birck R, Krzossok S, Markowetz F, Schnulle P, van der Woude FJ, Braun C. Acetylcysteine for prevention of contrast nephropathy: meta-analysis. Lancet. 2003 Aug 23;362(9384):598-603. doi: 10.1016/S0140-6736(03)14189-X. PMID 12944058
- [Background] Ward MM. Factors predictive of acute renal failure in rhabdomyolysis. Arch Intern Med. 1988 Jul;148(7):1553-7. PMID 3382301